CLINICAL TRIAL: NCT04962633
Title: Dietary Intervention With Probiotic Pasta and Evaluation of the Effects on Metabolic and Inflammatory Status in Overweight and Obese Subjects
Brief Title: Dietary Intervention With Probiotic Pasta and Evaluation of the Effects on Metabolic and Inflammatory Status
Acronym: ProPas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Paola Vitaglione, Associate Professor, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ProPas
Record Dates: First submitted 2021-06-10; First posted 2021-07-15 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic Pasta Group (Experimental): Subjects in the Probiotic Pasta group will consume 80 g per day of a probiotic pasta for 4 weeks
  Interventions: Other: Probiotic Pasta
- Control Pasta Group (Active Comparator): Control Pasta Subjects in the Control Pasta group will consume 80 g per day of conventional pasta for 4 weeks.
  Interventions: Other: Control Pasta

INTERVENTIONS:
Other: Probiotic Pasta — Subjects will consume for 4 weeks 80 g per day of probiotic durum wheat pasta. All subjects will be requested not to change the other daily dietary habits and their physical activity levels during the 4 week intervention period.
  Arms: Probiotic Pasta Group
Other: Control Pasta — Subjects will consume for 4 weeks 80 g per day of conventional durum wheat pasta without probiotics. All subjects will be requested not to change the other daily dietary habits and their physical activity levels during the 4 week intervention period.
  Arms: Control Pasta Group

SUMMARY:
This study aims to investigate the effects of daily consumption for 4 weeks of a probiotic durum wheat pasta vs a conventional durum wheat pasta without probiotics on fasting metabolic parameters and inflammatory status, on gut permeability and functionality, on daily energy intakes, appetite feelings, body weight, body mass index (BMI), waist and hip circumferences, blood pressure, body composition and wellbeing status in overweight and obese subjects.

DETAILED DESCRIPTION:
Growing evidence highlights the role of the individual diet and gut microbiome in modulating human metabolism, inflammatory status and cardiovascular risk.

This scenario supports nutritional approaches targeted to modify gut microbiota composition to trigger health benefits and the interest to develop novel functional foods enriched with probiotics. Most of commercial probiotic foods are in the category of dairy products and contain Lactobacillus strains. Besides that, Bacillus spp. along with the ability to form spores show probiotic attributes by exhibiting pathogen exclusion and antioxidant, antimicrobial and immune-modulatory abilities. Furthermore, they possess a stronger viability and stability to withstand high temperature processes, such as baking and boiling, than other probiotic bacteria thus representing an ideal choice for the development of functional cereal-based products.

In particular, Bacillus clausii UBBC07 exhibits probiotic properties by alleviating the severity and symptoms of acute diarrhoea in adults and children and show a high stability over a wide range of temperatures with potential applications in a variety of formulations and foods. The health benefits of B. clausii UBBC07 in overweight and obese subjects is unexplored.

This study aims to investigate the effects of consumption for 4 weeks of a probiotic durum wheat pasta enriched with spores of B. clausii UBBC07 vs a conventional durum wheat pasta (control) on metabolic and inflammatory status, on gut permeability and functionality, on daily energy intakes, appetite feelings, body weight, body mass index (BMI), waist and hip circumferences, blood pressure, body composition and wellbeing status in overweight and obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects;
* men and women;
* age 18-65 years;
* 25 kg/m2 ≤ BMI ≤ 35 kg/m2;
* habitual daily pasta consumption (≥ 1 portion/day);
* habitual diet characterized by absence of any food supplements and alternative medication, probiotics and prebiotics, whole grain and/or fiber enriched foods;
* intake of fruit/vegetables < 3 servings/day;
* low level of physical activity (< 500 metabolic equivalent min/week);
* signed written informed consent.

Exclusion Criteria:

* food allergies and intolerances and celiac disease;
* gastrointestinal diseases;
* relevant diseases;
* pregnant or breastfeeding;
* previous abdominal surgery;
* hypertriglyceridemia (Triglycerides > 200 mg/dL);
* hypercholesterolemia (Total cholesterol > 200 mg/dL);
* hyperglycaemia (glycaemia ≥ 110 mg/dL);
* hypertension (arterial blood pressure ≥140/90 mm Hg);
* weight loss ≥ 3 kg within 2 months before the study;
* antibiotics treatment within 3 months before the study;
* any medication (different from antibiotics) at the enrollment and within 2 months before the study;
* habitual diet characterized by high fruit and vegetables intakes (>3 portion/die);
* high level of physical activity;
* Alcohol consumption ≥ 3 alcohol units per day;
* simultaneous participation in other trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in fasting inflammatory blood markers | 1 months
  Measure of plasma C-reactive protein (mmol/L)
Changes in fasting plasma lipids | 1 months
  Measure of plasma concentrations (mg/dL) of Total-, LDL-, and HDL-Cholesterol, as well as Triglycerides
Changes in fasting plasma glucose | 1 months
  Measure of plasma glucose concentrations (mg/dL)

SECONDARY OUTCOMES:
Changes in small intestine permeability | 1 month
  Measure of lactulose and mannitol excreted in urines collected in the 0-5 hours time interval after an oral challenge with 5 g lactulose, 2 g mannitol and 2 g sucralose dissolved in 100 mL of water. The amounts of lactulose and mannitol excreted will be expressed in milligrams, and their ratio (lactulose/mannitol) will be calculated and used as marker of small intestine permeability
Changes in colonic permeability | 1 month
  Measure of sucralose excreted in urines collected over 24 hours after an oral challenge with 5 g lactulose, 2 g mannitol and 2 g sucralose dissolved in 100 mL of water. The amount of sucralose excreted will be expressed in milligrams and will be used as marker of colonic permeability
Changes in stool consistency | 1 month
  Measure of consistency of feces by mean of King's stool chart filled out by subjects. The chart comprises four categories of stool consistency: hard and formed, soft and formed, loose and unformed, liquid.
Changes in stool weight | 1 month
  Measure of stool weight by mean of King's stool chart filled out by subjects. The chart comprises three categories of stool weight : <100 g, 100-200 g, >200 g.
Changes in stool frequency | 1 month
  Measure of frequency of feces by mean of King's stool chart filled out by subjects. Fecal frequency is incorporated by recording the code of each feces passed over a 24 hour period.
Changes in gastrointestinal functionality | 1 month
  Calculation of daily fecal score from summation of all scores for stool consistency, weight and frequency obtained from King's stool chart filled out by subjects. Scores are weighted such that an increase in fecal frequency alone results in a higher score than a change in fecal consistency alone, which in turn results in a higher score than an increase in fecal weight alone. Diarrhea is classified by a daily fecal score of 15 or more.
Changes in faecal microbiome | 1 month
  The composition of faecal microbiome will be determined by high throughput sequencing of the 16S ribosomal ribonucleic acid (rRNA) gene. The massive number of sequences obtained will be analyzed by using state of the art bioinformatics tools and the presence and relative abundance of the microbial species occurring in each sample will be determined.
Variation of plasma glucagon like peptide-1 concentration | 1 month
  Measure of plasma glucagon like peptide-1 concentrations (mg/dL)
Variation of plasma gastric inhibitory polypeptide hormone concentration | 1 month
  Measure of plasma gastric inhibitory polypeptide concentrations (mg/dL)
Variation of plasma Glucagon hormone concentration | 1 month
  Measure of plasma Glucagon concentrations (mg/dL)
Variation of plasma Ghrelin hormone concentration | 1 month
  Measure of plasma Ghrelin concentrations (mg/dL)
Variation of plasma Insulin hormone concentration | 1 month
  Measure of plasma Insulin concentrations (mg/dL)
Variation of plasma endocannabinoids and N-acyl-ethanolamines concentration | 1 month
  Measure of plasma endocannabinoids and N-acyl-ethanolamines concentrations (mg/dL)
Variation of serum dipeptidyl-dipeptidase-IV activity | 1 month
  Measure of activity of dipeptidyl-dipeptidase-IV activity (U/L)
Changes in body weight | 1 month
  Measure of body weight in fasting subjects
Changes in body mass index | 1 month
  Calculation of body mass index by the formula weight in kilograms divided by height in meters squared.
Changes in waist circumference | 1 month
  Measure of waist circumference at the midpoint between the lower margin of the least palpable rib and the top of the iliac crest, with the tape parallel to the floor.
Changes in hip circumference | 1 month
  Measure of hip circumference around the widest portion of the buttocks, with the tape parallel to the floor.
Changes in blood pressure | 1 month
  Measure of systolic pressure and diastolic pressure in millimetres of mercury (mmHg) by using a digital sphygmomanometer
Changes in body composition | 1 month
  Body composition is determined by conventional bioelectrical impedance analysis with a single-frequency 50 kilohertz (kHz) bioelectrical impedance analyzer in the postabsorptive state (fasting subjects) and after being in the supine position for 20 min. Body composition data will be calculated from bioelectrical measurements and anthropometric data by using validated predictive equations.
Variation of daily energy intakes | 1 month
  Calculation of total daily energy intakes based on 7 days food records
Variation of hunger sensation scores | 1 month
  Measures of hunger sensation over the day reported by subjects by using hunger Visual Analogue Scales (VAS) 0-10 centimeters. Changes in these scores may reflect potential effects of dietary intervention in modulating hunger.
Variation of fullness sensation scores | 1 month
  Measure of fullness sensation over the day reported by subjects by using fullness Visual Analogue Scales (VAS) 0-10 centimeters. Changes in these scores may reflect potential effects of dietary intervention in modulating fullness.
Variation of satiety sensation scores | 1 month
  Measure of satiety sensation over the day reported by subjects by using satiety Visual Analogue Scales (VAS) 0-10 centimeters. Changes in these scores may reflect potential effects of dietary intervention in modulating satiety.
Variation of wellbeing status | 1 month
  Estimate of wellbeing status by mean of quality of life (QoL) questionnaire, which is based on Short Form-12 Health Survey (SF-12), a self-report form of subjective health. Physical and Mental Health Composite Scores (PCS & MCS) are computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.

CONTACTS AND LOCATIONS:
Overall Officials: Paola Vitaglione, Professor, Study Director — Department of Agricultural Sciences, Federico II University
Locations (1):
- Department of Agricultural Sciences, Portici, Italy

IPD SHARING:
Plan to Share IPD: Undecided
The investigators will decide as soon as data analysis are completed completed and there is a clear idea on publication rute according with the other coauthors.